CLINICAL TRIAL: NCT05249348
Title: A Phase 1 Open-label, Cross-over Study to Assess the Effects of Food on PC14586 Pharmacokinetics in Healthy Volunteers and to Assess PC14586 Pharmacokinetics in Healthy Japanese Volunteers Living in the US
Brief Title: Effect of Food on PC14586 in Healthy Volunteers and the PK of PC14586 in Healthy Japanese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PMV Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PMV-586-102; 262612 (Other: Parexel)
Record Dates: First submitted 2022-01-07; First posted 2022-02-21 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers
Keywords: Y220C; PC14586; PMV Pharma; PMV; food effect; Pharmacokinetics; Japanese

STUDY DESIGN:
Intervention Model Description: Single-dose crossover study one dose with food and one dose without food.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part 1 Sequence A (Experimental): Period 1 will be fed, then washout, then Period 2 will be fasted.
  Interventions: Drug: PC14586
- Part 1 Sequence B (Experimental): Period 1 will be fasted, then washout, then Period 2 will be fed.
  Interventions: Drug: PC14586
- Part 2 Sequence C (Experimental): Period 1 will be fed, then washout, then Period 2 will be fasted. A different dose of PC14586 will be tested.
  Interventions: Drug: PC14586
- Part 2 Sequence D (Experimental): Period 1 will be fasted, then washout, then Period 2 will be fed. A different dose of PC14586 will be tested.
  Interventions: Drug: PC14586
- Part 2 Japanese Cohort (Experimental): 6 Japanese participants will be administered a single dose of PC14586.
  Interventions: Drug: PC14586

INTERVENTIONS:
Drug: PC14586 — An oral dose of PC14586 will be used in Arms A and B (Part 1) and a different dose will be used for Arms C and D and the Japanese cohort (Part 2).

SUMMARY:
This is a 2-part Phase 1 cross-over study to assess the effects of food on the pharmacokinetics of PC14586 in healthy volunteers. The pharmacokinetics of PC14586 at a clinically relevant dose in Japanese participants will also be studied.

DETAILED DESCRIPTION:
PC14586 is a first-in-class, oral, small molecule p53 reactivator that is selective for the p53 Y220C mutation. This Phase 1 trial will be conducted in 2 parts (Part 1 - pilot and Part 2 - pivotal) to assess the pharmacokinetics of PC14586 in healthy volunteers including Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking male and female Caucasian/ non-Asian or Japanese human volunteers
* 18 to 55 years of age
* Able to swallow tablets.

Inclusion criteria for Japanese participants only:

* Japanese and born in Japan (1st generation)
* The parents and grandparents of the participant are ethnically Japanese and born in Japan
* Has undergone no significant change in lifestyle since leaving Japan
* Has lived < 10 years outside of Japan

Exclusion Criteria:

* Clinically significant medical history as determined by the PI.
* Any disorder that would interfere with the absorption, distribution, metabolism or excretion of drugs.
* A p53 Y220C mutation.
* Blood pressure >140 mm systolic or >90 diastolic.
* Smoked or used other nicotine-containing products during the previous 3 months.
* History of alcohol and/or illicit drug abuse within the previous 5 years.
* Hepatitis B surface antigen (HBsAg), Hepatitis C antibody or human immunodeficiency virus (HIV).
* Positive blood test for ethanol.
* Positive urine drug test.
* Pregnancy or breastfeeding.
* Unwilling to avoid use of alcohol or alcohol-containing foods, medications or beverages, within 48 hours prior to admission until discharge from the clinical site.
* Has donated blood within 2 months prior to admission.
* Has used over-the-counter (OTC) medications (including vitamins), prescription medications or herbal remedies from 14 days prior to admission.
* Has used an investigational drug within 30 days prior to Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Part 1: Effect of a high-fat meal on AUClast | 2 months
Part 1: Effect of a high-fat meal on AUC0-inf | 2 months
Part 1: Effect of a high-fat meal on the Tmax | 2 months
Part 1: Effect of a high-fat meal on the Cmax | 2 months
Part 2: Effect of a high-fat meal on the AUC0-last | 7 months
Part 2: Effect of a high-fat meal on the AUC0-inf | 7 months
Part 2: Effect of a high-fat meal on the Tmax | 7 months
Part 2: Effect of a high-fat meal on the Cmax | 7 months

SECONDARY OUTCOMES:
Part 1: Treatment emergent adverse events (TEAE) | 5 months
Part 1: Clinically relevant changes in: physical examinations, vital signs, clinical laboratory tests, 12-lead triplicate electrocardiogram (ECG) | 5 months
Part 2: AUC0-last of PC14586 | 6 months
Part 2: AUC0-inf of PC14586 | 6 months
Part 2: Cmax of PC14586 | 6 months
Part 2: Tmax of PC14586 | 6 months
Part 2: The apparent clearance (CL/F) of PC14586 | 6 months
Part 2: Volume of distribution (Vz/F) of PC14586 | 6 months
Half-life of PC14586 | 6 months
Part 2: Incidence of Treatment emergent adverse events (TEAE) | 10 months

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel Early Phase Clinical Unit - Los Angeles, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No